CLINICAL TRIAL: NCT00954876
Title: Phase II, Multi-Center, Open-Label, Prospective Study of Capecitabine and Cetuximab as First-Line Therapy in Patients With Metastatic Wild Type KRAS Colorectal Cancer Who Are Considered Nonoptimal Candidates or Are Intolerant to a First-Line Oxaliplatin/Irinotecan Regimen
Brief Title: Study of Capecitabine and Cetuximab as First-Line Therapy in Patients With Metastatic Wild Type Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: Translational Genomics Research Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-P02-07003
Record Dates: First submitted 2009-07-17; First posted 2009-08-07 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: capecitabine and cetuximab — Cetuximab 500 mg/m2 IV infusion over 1-2 hours Once every 2 weeks
  Capecitabine 1500 mg/m2 PO BID Days 1-7 followed by 7 days of no treatment and repeated every 2 weeks

SUMMARY:
The combination of capecitabine and cetuximab as first-line therapy will result in improved progression free survival compared to single agent capecitabine in patients with KRAS wild type colorectal cancer. Patients who are not able or willing to take Oxaliplatin/Irinotecan combination therapy are eligible for this study.

ELIGIBILITY:
Inclusion Criteria

* Metastatic colorectal cancer
* Tumor classified WT KRAS
* At least 18 yrs of age
* ECOG PS 0,1 or 2
* Evidence of adequate organ function
* Measurable disease per RECIST criteria
* Have at least two of the following criteria:

  * Age > 65 years
  * ECOG PS 1 or 2
  * Serum Albumin < or equal to 3.5g/dL
  * Prior RT to abdomen or pelvis
  * Stopped first-line combination systemic chemotherapy < 6 weeks duration

Exclusion Criteria

* Tumors classified as KRAS mutation
* Prior therapy with cetuximab, panitumumab or other agent that targets EGFR
* Prior exposure to any biologic
* Known sensitivity to cetuximab or 5-FU (or marked intolerance to 5-FU)
* Known DPD deficiency
* Uncontrolled angina or a myocardial infarction within the previous 12 months
* Concurrent severe uncontrolled medical illness
* Known uncontrolled CNS metastases
* Bowel disease associated with chronic diarrhea
* Major surgery within 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Primary objective is to assess PFS in patients with WT KRAS CRC treated with the combination regimen of capecitabine and cetuximab | 18 months

SECONDARY OUTCOMES:
To assess the response rate in patients with metastatic WT KRAS CRC treated with capecitabine and cetuximab | 18 months
To assess the overall survival rate among patients with metastatic WT KRAS CRC treated with capecitabine and cetuximab | 18 months
To characterize the toxic effects and AEs of the combination regimen of capecitabine and cetuximab in this patient population | every three months
To perform exploratory analyses of serum and tumor biomarkers (EGFR mutations and genotyping) on toxicity and efficacy. | 1 year after study closure

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Ramanathan, M.D., Principal Investigator — Translational Genomics
Locations (1):
- Evergreen Hematology & Oncology, Spokane, Washington, United States